CLINICAL TRIAL: NCT01770795
Title: A Phase II Trial of Genexol-PM and Gemcitabine in Patients With Advanced Non-small-cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Eun Kyung Cho, Professor, Gachon University Gil Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-GIRBA-2351
Record Dates: First submitted 2013-01-16; First posted 2013-01-18 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Non-small Cell Lung Cancer
Keywords: non-small cell lung cancer; gemcitabine; genexol-PM; paclitaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

ARMS (1):
- Genexol-PM/Gemcitabine (Experimental)
  Interventions: Drug: Genexol-PM/Gemcitabine

INTERVENTIONS:
Drug: Genexol-PM/Gemcitabine

SUMMARY:
To evaluate the efficacy and safety Genexol-PM(CrEL-free polymeric micelle formulated paclitaxel)and gemcitabine in untreated metastatic NSCLC patients

ELIGIBILITY:
Inclusion Criteria:

* age over 18
* histologically or cytologically confirmted non-small cell lung cancer
* stage IIIb with pleural effusion or stage IV
* ECOG PS 0-2
* at least one measurable lesion
* expected life span more than 3 months
* normal bone marrow, liver, renal function
* no prior chemotherapy or radiotherapy except for whole brain radiotherapy for symptomatic brain metastases
* more than 6 months from the last adjuvant chemotherapy

Exclusion Criteria:

* active infection
* severe comorbitidies
* pregnant or lactating women
* other invasive malignancies
* poorly controlled symptomatic brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2011-01; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Overall response rate | one year

SECONDARY OUTCOMES:
progression free survival | one year
overall survival | one year
toxicities | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Gachon University Gil Medical Center, Incheon, South Korea